CLINICAL TRIAL: NCT01559779
Title: The Effect of Gastric Bypass Surgery on the Beta- and Alpha Cells Secretory Function and the Insulinotropic Effect of the Incretin Hormones
Brief Title: Effect of Gastric Bypass Surgery on Pancreatic Islets and Incretin Function
Acronym: AB-CD-10
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Carsten Dirksen, MD PhD student, Hvidovre University Hospital
Other Study IDs: AB-CD-10
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
Keywords: Obesity; Roux-en-Y gastric bypass; Incretin hormones; Beta cell function
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum specimens are retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal glucose tolerance: Morbidly obese subjects with normal glucose tolerance undergoing gastric bypass surgery

SUMMARY:
The study aims at describing the acute and subacute changes after Roux-en-Y (RYGB) gastric bypass in insulin secretion from the beta cell and glucagon secretion from the alpha cell as well as the stimulatory effect of the incretins on the pancreatic islets. RYGB is a bariatric procedure that changes the gastrointestinal anatomy and has been demonstrated to cause remission of type 2 diabetes shortly after the operation, before any significant weight loss. The altered transit of nutrient through the gastrointestinal tract after the operation is thought to play a key role in this remission and studies have shown significant changes in the secretion of gut hormones, namely the incretin hormone glucagon-like peptide-1 (GLP-1). However it is unknown whether the secretory function of the pancreatic islets as well as the stimulatory effect of the incretin hormones is changes postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Normal glucose tolerance
* Age > 18 years
* BMI > 40 or > 35 if combined with hypertension or obstructive sleep apnoea
* Caucasian
* Normal hemoglobinaemia
* Signed informed consent

Exclusion Criteria:

* Major psychiatric disorder
* Alcohol or drug abuse
* Major hearth or pulmonary disease
* Previous major abdominal disease (e.g. peritonitis, large hernia)
* Pregnancy/lactation
* Treatment with GLP-1 analogs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from the population undergoing gastric bypass surgery at Hvidovre Hospital
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in beta cell function | Before and 1 week and 3 months after surgery
  Change in first and second phase insulin response, disposition index, and acute insulin secretion in response to a non-glucose stimulus
Insulinotropic effect of incretin hormones | Before and 1 week and 3 months after surgery
  Change in first and second phase insulin response during GLP-1 and GIP infusion compared to saline

SECONDARY OUTCOMES:
Change in alpha cell function | Before and 1 week and 3 months after surgery
  Change in glucagon secretion in response to glucose and non-glucose stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Dirksen, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Dpt. of Endocrinology (215) at Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Dirksen C, Bojsen-Moller KN, Jorgensen NB, Jacobsen SH, Kristiansen VB, Naver LS, Hansen DL, Worm D, Holst JJ, Madsbad S. Exaggerated release and preserved insulinotropic action of glucagon-like peptide-1 underlie insulin hypersecretion in glucose-tolerant individuals after Roux-en-Y gastric bypass. Diabetologia. 2013 Dec;56(12):2679-87. doi: 10.1007/s00125-013-3055-1. Epub 2013 Sep 19. PMID 24048673